CLINICAL TRIAL: NCT01108081
Title: An RCT of Telemedicine Interventions for OSA
Brief Title: Telemedicine Interventions for Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: IIR 09-063
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Sleep symptoms; Quality of Life
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): Physical activity
  Interventions: Behavioral: Physical activity
- Arm 2 (Experimental): Diet
  Interventions: Behavioral: Diet
- Arm 3 (Active Comparator): Health education
  Interventions: Behavioral: Health education
- Arm 4 (Experimental): Combined physical activity and diet
  Interventions: Behavioral: Physical activity; Behavioral: Diet

INTERVENTIONS:
Behavioral: Physical activity — Moderate-intensity physical activity
  Arms: Arm 1; Arm 4
Behavioral: Diet — Dietary weight loss
  Arms: Arm 2; Arm 4
Behavioral: Health education — Attention control intervention
  Arms: Arm 3

SUMMARY:
This project is investigating whether both moderate-intensity physical activity and dietary weight loss will independently reduce sleep apnea symptoms and improve quality of life.

DETAILED DESCRIPTION:
Background/Rationale:

Obstructive sleep apnea/hypopnea (OSAH) is a common chronic disease that is associated with daytime sleepiness, impaired health-related quality of life (QOL), and increased risk of hypertension and cardiovascular disease. The most common treatment is continuous positive airway pressure (CPAP), although adherence to CPAP is poor in more than one-third of patients. Weight loss can clearly lessen the severity of OSAH, but although short-term dietary weight loss can often be achieved it is difficult to maintain. Regular aerobic exercise is associated with a lower prevalence of OSAH in observational studies after adjustment for body habitus, and in two small clinical trials moderate exercise was associated with a substantial decrease in OSAH severity despite little or no weight loss. Demonstrating that dietary weight loss and moderate physical activity, promoted in the home setting, independently improve OSAH severity will have a major impact on the therapeutic approach to OSAH, a disease that is highly prevalent in the VA population.

Objective:

The investigators hypothesize that both moderate-intensity physical activity and dietary weight loss will independently reduce OSAH severity and improve QOL.

Methods:

The proposed study is a randomized clinical trial designed to test the independent effects of the physical activity and diet interventions, with an attention control intervention for subjects not assigned to either active intervention. Subjects will be male and female Veterans with a BMI over 24 kg/m2, with a physician diagnosis of OSAH and apnea-hypopnea index (AHI) >10/hr. The interventions will last six months.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of sleep apnea
* Apnea-hypopnea index >10/hr
* BMI over 24 kg/m2

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-10; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity: Physical activity
  Physical activity: Moderate-intensity physical activity
- Diet: Diet
  Diet: Dietary weight loss
- Health Education: Health education
  Health education: Attention control intervention
- Combined Physical Activity/Diet: Combined physical activity and diet
Period: Overall Study
Arm/Group | Physical Activity | Diet | Health Education | Combined Physical Activity/Diet
Started | 46 | 42 | 38 | 43
Completed | 44 | 40 | 38 | 39
Not Completed | 2 | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity | Diet | Health Education | Combined Physical Activity/Diet | Total
Number analyzed (Participants) | 46 | 42 | 38 | 43 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0) | 60.5 (8.7) | 59.1 (11.0) | 56.3 (10.0) | 59.5 (9.8)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 3 | 5
  Male | 44 | 42 | 38 | 40 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change Over 6 Months in Epworth Sleepiness Scale Score
Description: Epworth Sleepiness Scale score, change in score from baseline to 6 months. Total scores range from 0-24, where higher scores indicate more sleepiness.
Time Frame: baseline and 6 months
Population: Two participants did not complete the questionnaire and therefore had missing Epworth Sleepiness Scale scores. One participant in Diet arm and one participant in Health education arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physical Activity | Diet | Health Education | Combined Physical Activity/Diet
Number analyzed (Participants) | 44 | 39 | 37 | 39
units on a scale | -0.23 (0.69) | -1.05 (0.38) | 0.43 (0.66) | -2.62 (0.59)

2. Secondary Outcome: Change Over 6 Months in Quality of Life
Description: Quality of life as assessed by the Functional Outcomes of Sleep Questionnaire, change from baseline to 6 months. The potential range of scores for the Functional Outcomes of Sleep total score is 5-20 where higher scores indicate better quality of life. The total score is the sum of the 5 subscale scores (general productivity, social outcome, activity level, vigilance, intimate relationships), which are weighted means ranging from 1-4.
Time Frame: baseline and 6 months
Population: Two participants did not complete the questionnaire and therefore had missing Functional Outcomes of Sleep Questionnaire scores. One participant in Diet arm and one participant in Health education arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physical Activity | Diet | Health Education | Combined Physical Activity/Diet
Number analyzed (Participants) | 44 | 39 | 37 | 39
units on a scale | 0.24 (0.44) | 0.15 (0.24) | -0.33 (0.28) | 1.24 (0.42)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Physical Activity | Diet | Health Education | Combined Physical Activity/Diet
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/42 | 0/38 | 0/43
Other Adverse Events (participants affected / at risk) | 0/46 | 0/42 | 0/38 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes